CLINICAL TRIAL: NCT06750302
Title: The Effectiveness of Inhaled Methoxyflurane (Penthrox) vs Placebo for Pain Relief in Coblation and Sinus Procedures: a Double-blind, Randomized, Placebo - Controlled Trial
Brief Title: Effectiveness of Penthrox vs Placebo in Sinus Procedures, a Clinical Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Director, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H24-02351
Record Dates: First submitted 2024-11-29; First posted 2024-12-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-12

CONDITIONS: Chronic Rhinosinusitis (CRS)
Keywords: Chronic Rhinosinusitis (CRS); Sinus Surgery; Endoscopic Sinus Surgery (ESS); Coblation; Methoxyflurane; Penthrox; Inhaled Analgesic; Inhaled Analgesics in Rhinology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Penthrox (Active Comparator): 3mL Penthrox as an inhaled analgesic
  Interventions: Drug: Methoxyflurane - Penthrox
- Placebo (Placebo Comparator): 3mL placebo control (saline + one drop of methoxyflurane)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methoxyflurane - Penthrox — 3ml
  Arms: Penthrox
Other: Placebo — saline + one drop of methoxyflurane
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effectiveness of inhaled methoxyflurane (Penthrox) as an analgesic for patients undergoing minor rhinology and sinus procedures, specifically comparing it to a placebo control. The primary question the study aims to answer is:

Does methoxyflurane provide superior pain relief compared to placebo during minor sinus procedures, as measured by the Visual Analog Scale (VAS)? If there is a comparison group: Researchers will compare the effects of Penthrox to the placebo (saline + one drop of methoxyflurane) to see if it provides better pain relief, reduces anxiety, and leads to fewer complications, including bleeding.

Participants will be asked to:

Inhale 3 mL of Penthrox or placebo during their procedure. Complete a VAS scale to assess pain. Complete anxiety assessments pre- and post-operatively. Be monitored for complications such as bleeding and other adverse effects. This study will help determine the effectiveness of Penthrox as a non-invasive, quick-acting analgesic for minor sinus surgeries.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled trial aims to assess the efficacy of methoxyflurane (Penthrox) as an inhaled analgesic for patients undergoing minor sinus and rhinology procedures, specifically sinus surgery and coblation procedures, compared to a placebo control.

Background and Rationale Sinus surgery, including procedures such as Endoscopic Sinus Surgery (ESS) and coblation (a type of surgical ablation), is commonly performed to treat chronic rhinosinusitis (CRS), sinus obstruction, and other sinus-related conditions. However, many of these procedures, especially those conducted in the office setting, require the use of local anesthesia for pain control. Current methods of pain management, such as local anesthetic injections (e.g., lidocaine, bupivacaine), are effective but can cause anxiety and discomfort for patients, especially when multiple injections are needed. Thus, there is a significant need for a more comfortable, non-invasive, and efficient analgesic approach to improve patient experience during these procedures.

Methoxyflurane (Penthrox) is an inhaled analgesic that has been widely used in Australia and New Zealand for trauma-related pain management for over 30 years and was approved for use in Canada in 2018. It is a short-acting, inhaled analgesic with a rapid onset of action and has shown promising results in treating acute pain in emergency and trauma settings. However, limited studies have explored its use in minor surgical procedures, particularly in the field of otolaryngology. Preliminary data from studies in other surgical disciplines, such as urology, suggest that methoxyflurane can provide effective analgesia in office-based procedures, with minimal side effects. This trial seeks to expand this body of evidence by evaluating Penthrox as an alternative to local anesthetic injections in sinus and rhinology surgeries.

Study Design This is a double-blind, parallel-arm, randomized controlled trial designed to assess the analgesic efficacy of Penthrox in patients undergoing minor sinus procedures, including sinus surgery and coblation, compared to a placebo control.

Primary Hypothesis: Inhaled methoxyflurane will provide superior pain relief during and after the procedure compared to the placebo, as measured by Visual Analog Scale (VAS) for pain.

Secondary Hypotheses: Methoxyflurane will reduce anxiety (measured by the APAIS score) and be associated with fewer complications (e.g., bleeding, adverse events) compared to placebo.

A total of 100 patients will be enrolled in the study, with 50 patients per group. The patients will be randomized into two arms: one receiving 3 mL of methoxyflurane and the other receiving 3 mL of placebo (saline + one drop of methoxyflurane to mimic the smell of the active drug, ensuring proper blinding).

Randomization will be stratified based on the type of procedure (i.e., coblation or sinus surgery) to ensure an even distribution of participants across the groups. Block randomization will be used to allocate patients to one of the two groups, with varying block sizes of 2-6 to maintain allocation concealment. The patient and surgeon will be blinded to the treatment allocation to minimize bias in assessment and administration.

Study Procedures and Interventions Inhalation of Methoxyflurane: Participants in the treatment group will inhale 3 mL of methoxyflurane (Penthrox) through a self-administered inhaler device immediately before and during their procedure. The inhaler is designed to deliver the appropriate concentration of methoxyflurane, providing rapid onset analgesia.

Inhalation of Placebo: Participants in the control group will inhale 3 mL of a placebo solution, which consists of saline with one drop of methoxyflurane to simulate the smell of the active drug. This is designed to maintain the blinding of the study.

The analgesic effect will be assessed during the procedure and at multiple time points post-operatively using the Visual Analog Scale (VAS). Anxiety levels will be measured using the APAIS score before and after the procedure. Surgical complications such as bleeding, pain, and adverse reactions will be monitored throughout the procedure.

Primary Outcome Measures VAS Score: The primary endpoint for the study will be the patient-reported pain score using a Visual Analog Scale (VAS), which measures the intensity of pain during the procedure and for a period of time after the procedure (e.g., 1 hour, 24 hours, and 1 week post-op).

Pain Characteristics: In addition to VAS, other pain characteristics will be assessed, including pain duration, frequency, and any additional pain management required during the procedure.

Secondary Outcome Measures Type of Procedure: An analysis of whether the analgesic effect differs between procedures (i.e., coblation vs. sinus surgery).

SNOT-22 Scores: Pre- and post-operative SNOT-22 scores will be collected at 4, 8, and 12 weeks to assess the effect of the procedure and analgesic treatment on sinus symptoms and quality of life.

Bleeding and Adverse Events: The occurrence of any surgical complications (e.g., bleeding, infection) or adverse effects (e.g., nausea, dizziness) will be closely monitored during and after the procedure.

Anxiety Levels: Anxiety will be assessed using the APAIS (Anxiety and Pain Assessment Index) before and after the procedure to determine the impact of Penthrox on patient anxiety.

Statistical Analysis Data analysis will compare the pain scores, surgical outcomes, and adverse events between the treatment and placebo groups. Primary analysis will focus on the VAS scores at different time points. Secondary analyses will compare differences in anxiety, complications, and post-operative recovery. A stratified analysis will be performed based on procedure type (coblation vs. sinus surgery).

Safety and Monitoring The study will be conducted under strict adherence to Good Clinical Practice (GCP) guidelines. Safety monitoring will be performed by a designated safety officer, and any serious adverse events (SAEs) will be reported to the study coordinator and the regulatory authorities as required. Participants will receive appropriate care for any complications, and the study will be paused or terminated if safety concerns arise.

Ethical Considerations This study has been designed to ensure the safety and wellbeing of all participants. All participants will provide informed consent before enrollment, and their participation will be voluntary. The study protocol has been reviewed and approved by a recognized ethics review board.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Scheduled for minor sinus surgery or coblation procedures

Exclusion Criteria:

* Cystic fibrosis
* Systemic vasculitis or other bleeding disorders
* History of renal failure or severe kidney disease
* History of liver failure or severe liver disease
* Altered state of consciousness (head injury, alcohol use, drug use)
* Known or suspected hypersensitivity to lidocaine or sensorcaine
* Inhaled drug use (i.e., cocaine) in the preceding 6 months
* Nasal tumors
* Personal or family history of malignant hyperthermia
* Respiratory depression

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-24 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for Pain | Immediately post-procedure, 1 hour post-procedure, and at 24 hours post-procedure.
  This scale measures the intensity of pain experienced by the participant during and immediately after the procedure. Participants will rate their pain on a scale from 0 (no pain) to 10 (worst pain imaginable) at various time points: immediately post-procedure, 1 hour post-procedure, and at 24 hours post-procedure. The primary goal is to compare the pain relief provided by methoxyflurane (Penthrox) versus the placebo.
Pain Duration | It will be recorded as the time (in minutes or hours) from the end of the procedure until the participant reports no significant pain in a time frame of 4 hours
  This measure tracks the duration of pain experienced by the participant post-surgery. This will help assess how long the pain relief from methoxyflurane lasts compared to the placebo.
Numeric Pain Rating Scale (NPRS) | Immediately post-procedure, 1 hour post-procedure, and at 24 hours post-procedure.
  The NPRS will be used as a secondary assessment to quantify the severity of pain. Patients will rate their pain on a scale from 0 to 10, with 0 being no pain and 10 being the worst pain imaginable. The NPRS is a simpler and widely used scale for self-reported pain.
Amount of Local Anesthetic Injections | Immediately post-procedure, 1 hour post-procedure, and at 24 hours post-procedure.
  his outcome measures the total number of local anesthetic injections (e.g., lidocaine or bupivacaine) required during the procedure. Fewer injections may indicate better pain control with the study intervention (methoxyflurane) as compared to the placebo. This will help assess the need for additional pain management during surgery.
Patient Perception of Analgesic Effect | Immediately post-procedure, 1 hour post-procedure, and at 24 hours post-procedure.
  After the procedure, participants will be asked to report their perception of pain relief and whether they felt the analgesic effect was sufficient during the procedure. The outcome will be assessed through a self-reported survey where participants rate the effectiveness of the pain management on a Likert scale (e.g., from very effective to not effective at all).

SECONDARY OUTCOMES:
Type of Procedure | At surgery time
  This measure records the specific type of minor sinus procedure the participant undergoes (e.g., coblation procedure or sinus surgery). This is important because different procedures may have varying levels of pain and complication risk, and it allows the study to analyze if the effectiveness of methoxyflurane varies based on the type of procedure.
Field of View During Surgery | At surgery time
  The field of view refers to the surgeon's ability to see and access the surgical site during the procedure, which could be affected by pain, swelling, or bleeding. This will be assessed by the surgeon and recorded for both treatment groups to help determine if methoxyflurane has an impact on the ease or quality of the procedure.
Estimated Blood Loss in milliliters | At surgery time
  This outcome measures the amount of blood lost during the procedure. It's particularly relevant for sinus surgeries, as excessive bleeding can affect the success of the surgery and recovery. Lower blood loss may be associated with better procedural conditions, potentially influenced by the use of methoxyflurane for pain management and sedation.
SNOT-22 Score | It will be administered pre-operatively, as well as at 4, 8, and 12 weeks post-op
  The SNOT-22 (Sinusitis Symptom Scale) is a widely used questionnaire assessing the severity of sinus-related symptoms, such as nasal congestion, facial pain, loss of smell, and overall quality of life.
APAIS Score (Anxiety and Pain Assessment) | Pre-operative
  The APAIS (Amsterdam Preoperative Anxiety and Information Scale) is a tool used to assess anxiety levels in patients prior to the procedure. This will be measured pre-operatively and compared between groups to determine whether methoxyflurane provides any anxiolytic (anti-anxiety) effects compared to the placebo.
Anxiety Levels During and Post-Operative (Likert scale) | Pre-operative (1 hour) and Post-operative (up to 4 hours)
  Anxiety will be assessed using a self-reported scale during the procedure (if feasible, based on patient condition) and post-operatively. Participants will rate their anxiety on a Likert scale, allowing the study to determine whether methoxyflurane has an anti-anxiety effect in addition to its analgesic properties. Post-operative anxiety is especially important, as it may influence recovery and patient satisfaction.
Adverse Events | Immediately post-procedure, 1 hour post-procedure, and at 24 hours post-procedure.
  Adverse events and complications (e.g., bleeding, infection, other procedural issues) that occur during or after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- St Paul's Sinus Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No